CLINICAL TRIAL: NCT05340712
Title: Evaluation of the Efficacy of a New Specific Infant Formula With a Prebiotic and Probiotics in Case of Functional Constipation
Brief Title: Evaluation of the Efficacy of a New Specific Infant Formula in Case of Functional Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United Pharmaceuticals (Industry)
Collaborators: Delta Consultants (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UP2021-02-FALCON
Record Dates: First submitted 2022-04-08; First posted 2022-04-22 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Functional Constipation
Keywords: Constipation; Infants; Infant formula; Nutrition; Defecation; Prebiotic; Probiotics
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Superiority, double-blind, randomized, placebo-controlled trial of 60 days followed by an optional 60 day, open-label follow-up period with the tested formula only
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation of the formula to each infant is drawn according to a randomization list developed using a software by the clinical research organization in charge of statistics and known only to him until the blind is lifted, i.e. after the statistical analysis. A 1:1 double-blind randomisation will be computer-generated by block (in each center).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IT formula (Experimental): The test product (IT formula) is an infant formula based on cow's milk proteins containing a high level of lactose, a prebiotic, a high concentration of magnesium and a mix of probiotics.
  Interventions: Dietary Supplement: new infant formula
- Standard formula (Placebo Comparator): The control product is a standard infant formula based on cow's milk proteins containing usual lactose and magnesium content, no prebiotic nor probiotic.
  Interventions: Dietary Supplement: Standard formula

INTERVENTIONS:
Dietary Supplement: new infant formula — New formula containing a prebiotic and a mix of probiotics, randomly assigned to infants during a 2-month period and allocated to all infants during the optional open-label follow-up period of 2 months.
  Arms: IT formula
Dietary Supplement: Standard formula — Standard infant formula containing no prebiotic nor probiotic, randomly assigned to infants during a 2-month period followed by an optional open-label follow-up period of 2 months with the new infant formula
  Other Names: Novalac 1
  Arms: Standard formula

SUMMARY:
This study aims to assess the clinical efficacy, safety and tolerance of a new formula containing a prebiotic and a mix of probiotics in the specific population of infants suffering from functional constipation through a superiority, double-blind, randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
The study comprises a selection period of 1 week where the eligibility of the infant to participate in the study will be evaluated. Once his/her participation is confirmed, the tested formula will be compared to a standard formula during a 2-month study period followed by an optional follow-up period of 2 months where only the tested formula will be used.

ELIGIBILITY:
Selection Criteria:

Infants presenting with constipation according to modified Rome IV criteria, i.e. they must present with 1 month the following:

* Infants without spontaneous stools or with at least one painful or hard spontaneous bowel movement per week AND
* At least one of the following:

  * Two and fewer spontaneous defecations per week
  * History of excessive stool retention
  * History of large-diameter stools

Non-selection Criteria (non-exhaustive list):

* Preterm birth (<34 weeks of gestational age)
* Exclusively or partially breastfed infants within 3 days prior to visit V-1
* Infants with organic causes of constipation (e.g. coeliac disease, paediatric intestinal pseudo-obstruction, hypothyroidism, spina bifida, anorectal malformation or Hirschsprung's disease) or constipation secondary to endocrine, metabolic, neurologic or autoimmune disorders, surgery or drugs.
* Infants on laxative treatment
* Infants taking drugs that are known to affect gastrointestinal motility as well as any probiotic supplements
* Infants treated with antibiotics
* Infants with a known allergy to one of the formula ingredients (e.g. cow's milk proteins…)
* Infants with anaemia who have been prescribed an oral iron supplement as treatment
* Infants participating in another trial
* Infants presenting with any other situation which, according to the investigator, may interfere with the study participation, or lead to a particular risk for the infant

Inclusion Criteria:

* Infants having completed the selection period and still compliant with non-selection criteria
* Infants being constipated according to modified Rome IV criteria based on information recorded in parents' diary during the week preceding visit V0 (inclusion visit)

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Hard stool consistency or painful defecation | 30 days
  Proportion of hard or painful stools per total number of spontaneous bowel movements by participant. A spontaneous bowel movement is defined as described in outcome 2.
  Stool consistency will be evaluated based on the Brussels Infant and Toddler Stool Scale (BITSS). BITSS is a reliable instrument to assess stools of non-toilet trained children. It consists of color photographs of nappies containing stools from infants and toddlers categorized as hard, formed, loose, or watery (Huysentruyt et al., 2019).
  The consistency and painful defecation of each stool will be assessed by parents at Day 30.

SECONDARY OUTCOMES:
Total and spontaneous defecation frequency | 30, 60, 90 and 120 days
  Spontaneous bowel movement is defined as a bowel movement not produced by the use of rescue medication. Stools occurring within 24h after the use of rescue medication will not be considered spontaneous. If 2 stools occur within less than 1 hour, only 1 stool will be considered (Koppen et al., 2018).
  Defecation frequency will be assessed by parents by recording the time of each stool during the week preceding each visit.
Stool consistency | 30, 60, 90 and 120 days
  Parents will record the consistency of every stool the week preceding each visit as described in the outcome 1 using the BITSS scale (Brussels Infant and Toddler Stool Scale) which consists of 4 stools consistency categories (hard, formed, loose, or watery ; Huysentruyt et al., 2019)
Painful defecation | 30, 60, 90 and 120 days
  Painful defecation will be evaluated by parents for each stool during the week preceding each visit (Yes/No).
Excessive stool retention | 30, 60, 90 and 120 days
  "Excessive stool retention" is defined as "the infant withholding stools". It will be evaluated by parents at each visit (presence/absence).
Large diameter stools | 30, 60, 90 and 120 days
  Large diameter stools will be assessed by parents at each visit using the picture of the largest stool in the BITSS as an example of the large diameter stool (presence/absence).
Treatment success | 30, 60, 90 and 120 days
  Treatment success is defined as no longer meeting the modified Rome IV criteria for functional constipation, i.e. the treatment will be considered as a success if the infant does not meet more than one of the following criteria per week during the week preceding each visit:
  1. At least one painful or hard spontaneous bowel movement (Yes/No)
  2. Two or fewer spontaneous defecations per week (Yes/No)
  3. Excessive stool retention (Yes/No)
  4. Large-diameter stools (assessed using the BITSS as described in the outcome 6) (Yes/No)
Rescue medication use | 30, 60, 90 and 120 days
  The frequency of use, type and dosage of rescue medication will be assessed by parents during the whole study.
Weight | 30, 60, 90 and 120 days
  Weight will be expressed in kg and in z scores according to the World Health Organization (WHO) Child Growth Standards.
Height | 30, 60, 90 and 120 days
  Height will be expressed in cm and in z scores according to the WHO Child Growth Standards.
Head circumference | 30, 60, 90 and 120 days
  Head circumference will be expressed in cm and in z scores according to the WHO Child Growth Standards.
BMI | 30, 60, 90 and 120 days
  BMI will be expressed in value and z scores according to the WHO Child Growth Standards.
Adverse events | Through study completion, i.e. 67 days or 127 days if participation to the optional follow-up period
  Any untoward medical condition occurring during the study in an infant receiving study products regardless of a causal relationship with the product or not will be considered an adverse event and reported as such. This definition includes events occurring from the moment the parents have signed the Informed Consent form (day -7) up until the study end (or early termination).
Nutritional status | 0 and 60 days
  Nutritional status will be assessed based on the evaluation of specific blood biological markers (albumin, creatinine, urea, hemoglobin, sodium, potassium, chloride).
Crying time | 30, 60, 90 and 120 days
  Daily crying duration will be assessed by parents on 3 days in the week preceding each visit.
Regurgitations | 30, 60, 90 and 120 days
  The number of regurgitation episodes, the volume of regurgitation and regurgitation severity will be assessed by parents on 3 days in the week preceding each visit. Regurgitation severity will be assessed through the Vandenplas score ranging from 0 (=less than 2 regurgitation episodes / day) to 6 (=regurgitation of the complete volume after each feeding).
Sleep quality | 30, 60, 90 and 120 days
  Sleep quality will be evaluated by parents at each visit by asking them if their child's sleep was quiet or agitated.
Sleep time satisfaction | 30, 60, 90 and 120 days
  Sleep time satisfaction will be evaluated by parents at each visit (Yes/No).
Parents' quality of life (QoL) | 30, 60, 90 and 120 days
  Parents' QoL will be assessed based on a questionnaire adapted from the Parental Opinions of Pediatric Constipation (POOPC) scale (Silverman et al., 2015). Questions from this scale were chosen based on their relevance to constipated infants. This questionnaire is composed of 4 items, i.e. Burden/Worry, Family, Treatment and Social. Each question is scored on a scale of 1 (=Strongly Disagree) to 5 (=Strongly Agree) with higher scores indicating that infant's constipation greatly affects parents' QoL. The total score is calculated by summing the scores of all individual question, ranging from 15 to 75 where a score of 15 indicates that infant's constipation does not affect parents' QoL whereas a score of 75 indicates that parents' QoL is extremely affected by infant's constipation.
Parents' satisfaction | 30, 60, 90 and 120 days
  Parents' adequate relief will be assessed at each visit (Yes/No).
Gut microbiota composition | 0 and 60 days
  Gut microbiota composition will be analyzed by 16S rRNA gene sequencing from stool samples.
Short-chain fatty acids (SCFAs) | 0 and 60 days
  SCFAs will be measured in stool samples by gas chromatography/mass spectrometry (GC/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Staiano, Prof., Study Director — Federico II University; Marc Benninga, Prof., Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Caterina Strisciuglio, Prof., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (2):
- Italy (2):
  - University of Naples "Federico II", Napoli
  - University of Campania Luigi Vanvitelli, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huysentruyt K, Koppen I, Benninga M, Cattaert T, Cheng J, De Geyter C, Faure C, Gottrand F, Hegar B, Hojsak I, Miqdady M, Osatakul S, Ribes-Koninckx C, Salvatore S, Saps M, Shamir R, Staiano A, Szajewska H, Vieira M, Vandenplas Y; BITSS working group. The Brussels Infant and Toddler Stool Scale: A Study on Interobserver Reliability. J Pediatr Gastroenterol Nutr. 2019 Feb;68(2):207-213. doi: 10.1097/MPG.0000000000002153. PMID 30672767
- [Background] Koppen IJN, Saps M, Lavigne JV, Nurko S, Taminiau JAJM, Di Lorenzo C, Benninga MA. Recommendations for pharmacological clinical trials in children with functional constipation: The Rome foundation pediatric subcommittee on clinical trials. Neurogastroenterol Motil. 2018 Apr;30(4):e13294. doi: 10.1111/nmo.13294. Epub 2018 Jan 30. PMID 29380480
- [Background] Silverman AH, Berlin KS, Di Lorenzo C, Nurko S, Kamody RC, Ponnambalam A, Mugie S, Gorges C, Sanghavi R, Sood MR. Measuring Health-Related Quality of Life With the Parental Opinions of Pediatric Constipation Questionnaire. J Pediatr Psychol. 2015 Sep;40(8):814-24. doi: 10.1093/jpepsy/jsv028. Epub 2015 Apr 2. PMID 25840448